CLINICAL TRIAL: NCT03794362
Title: Developing a Method to Objectively Measure Analgesic Interventions: A Pilot Study
Brief Title: Measuring Analgesic Interventions
Status: Recruiting | Type: Observational
Sponsor: Julia Finkel (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 9586
Record Dates: First submitted 2018-10-31; First posted 2019-01-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: analgesia; pain; nociception; pupillometry; analgesic
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (6):
- Local Anesthetics: Lidocaine
- N-methyl-D-aspartate Antagonists: Ketamine
- SNRIs: Duloxetine
- Alpha-2 adrenergic agonists: Dexmedetomidine
- Oral Analgesics: NSAIDs, acetaminophen
- Non-pharmacologic interventions: Acupuncture

SUMMARY:
It is generally recognized that pain assessment and management especially in newborns, children and other nonverbal populations is an unmet need. According to the American Medical Association, "the pediatric population is at risk of inadequate pain management, with age-related factors affecting pain management in children. Children are often given minimal or no analgesia for procedures that would routinely be treated aggressively in adults. Although much is now known about pain management in children, it has not been widely or effectively translated into routine clinical practice". These two factors combine to emphasize the necessity for an objective tool to quantify pain and monitor the effectiveness of analgesia, especially during treatments. Further, it is reported that many patients require a combination of treatments, and it is often necessary to test a variety of treatments before the personal match for treatment is found. The method in place to change the care on a subjective basis is difficult, time consuming, and not easily individualized. This pilot study is part of an ongoing effort to develop a method to objectively assess response to specific analgesic interventions. It specifically aims to discern the impact of analgesic interventions on sensory nerve fiber sensitivity in a diverse patient population.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 7 to 21 years of age
2. The subject is receiving an analgesic intervention in the Children's National Medical Center Pain Clinic
3. The subject is willing and able to provide written informed assent/parental consent to the study participation.

Exclusion Criteria:

1. Eye pathology precluding pupillometry
2. Patients who are actively using opioids (history of use acceptable). Rationale: opioids constrict the pupil, and therefore concomitant opioid use would bias our results.
3. Subjects who are or may be pregnant

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are receiving pharmacological or non-pharmacological analgesic interventions as part of their regularly occurring clinical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pupillary Reflex Dilation (PRD) Area under Curve (AUC) | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The changes that occur in PRD AUC as a response to an analgesic intervention will be investigated. The differences are calculated by comparing the parameters from before the intervention to after the intervention.

SECONDARY OUTCOMES:
Pupillary Light Reflex (PLR) Latency | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The changes that occur in PLR Latency as a response to an analgesic intervention will be investigated. The differences are calculated by comparing the parameters from before the intervention to after the intervention.
Pupillary Light Reflex (PLR) Amplitude | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The changes that occur in PLR Amplitude as a response to an analgesic intervention will be investigated. The differences are calculated by comparing the parameters from before the intervention to after the intervention.
Pupillary Light Reflex (PLR) Recovery Time | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The changes that occur in PLR Recovery Time as a response to an analgesic intervention will be investigated. The differences are calculated by comparing the parameters from before the intervention to after the intervention.
Pupillary Reflex Dilation (PRD) Amplitude | 0, 15, 30, 45, 60, 90, 120, 180 minutes
  The changes that occur in PRD amplitude as a response to an analgesic intervention will be investigated. The differences are calculated by comparing the parameters from before the intervention to after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States